CLINICAL TRIAL: NCT04591431
Title: The Rome Trial From Histology to Target: the Road to Personalize Target Therapy and Immunotherapy
Acronym: ROME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione per la Medicina Personalizzata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR-BAS-18-005; 2018-002190-21 (EudraCT Number)
Record Dates: First submitted 2020-09-18; First posted 2020-10-19 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Gastrointestinal Cancer; Non Small Cell Lung Cancer; Other Cancer
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Trastuzumab; Ado-Trastuzumab Emtansine; pertuzumab; Lapatinib; Everolimus; Vemurafenib; cobimetinib; alectinib; brigatinib; palbociclib; ponatinib; itacitinib; ipatasertib; entrectinib; atezolizumab; Nivolumab; Ipilimumab; pemigatinib; pralsetinib; selpercatinib; talazoparib; tepotinib; Alpelisib

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, multicenter, Proof of Concept, Phase II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored Therapy (Experimental): Experimental (TT) Patients will be treated with target therapy and/or immunotherapy according to their genomic profile evidenced by Foundation One test and independently from their type of cancer with one or more drugs of the following list (administered according to the SmPCs or IBs if under development):
  TARGET THERAPY: ERLOTINIB (EGFR mutation) TRASTUZUMAB, PERTUZUMAB, TDM1, LAPATINIB (ERBB2 amplifications/mut) EVEROLIMUS (mTOR mutations, AKT mut) VEMURAFENIB, COBIMETINIB (BRAFV600E mutations) ALECTINIB, BRIGATINIB (ALK, RET) PALBOCICLIB (CDK4/6, CDKN2A/p16) PONATINIB (Bcr-abl) VISMODEGIB (SMO/PTCH1) ITACITINIB (JAK mutation) INCB054828 (FGFR1/2/3) IPATASERTIB (PI3K, AKT, PTEN) ENTRECTINIB (NTRK1/2/3 -TRK fusion proteins-, ROS1) ALPELISIB (PI3K, AKT) TEPOTINIB (MET amplification/exon14 skipping mutations) PRALSETINIB (RET) TALAZOPARIB (BRCA1/2, ATM, other HRD status) SELPERCATINIB (RET) IMMUNOTHERAPY: ATEZOLIZUMAB, NIVOLUMAB, IPILIMUMAB (MSI, HIGH TUMOR MUTATIONAL BURDEN, OTHER)
  Interventions: Drug: Erlotinib; Drug: Trastuzumab; Drug: Trastuzumab emtansine; Drug: Pertuzumab; Drug: Lapatinib; Drug: Everolimus; Drug: Vemurafenib; Drug: Cobimetinib; Drug: Alectinib; Drug: Brigatinib; Drug: Palbociclib; Drug: Ponatinib; Drug: Vismogedib; Drug: Itacitinib; Drug: Ipatasertib; Drug: Entrectinib; Drug: Atezolizumab; Drug: Nivolumab; Drug: Ipilimumab; Drug: Pemigatinib; Drug: Pralsetinib; Drug: Selpercatinib; Drug: Talazoparib; Drug: Tepotinib; Drug: Alpelisib
- Standard of Care (Active Comparator): Patients will be treated according the current version of the AIOM (Italian Association of Medical Oncology) guidelines for their type of cancer. As an example, patients could be treated with standard chemotherapy and/or targeted therapy according to the histological results.
  Interventions: Drug: Oncology Drugs

INTERVENTIONS:
Drug: Erlotinib — TT arm
  Arms: Tailored Therapy
Drug: Trastuzumab — TT arm
  Arms: Tailored Therapy
Drug: Trastuzumab emtansine — TT arm
  Arms: Tailored Therapy
Drug: Pertuzumab — TT arm
  Arms: Tailored Therapy
Drug: Lapatinib — TT arm
  Arms: Tailored Therapy
Drug: Everolimus — TT arm
  Arms: Tailored Therapy
Drug: Vemurafenib — TT arm
  Arms: Tailored Therapy
Drug: Cobimetinib — TT arm
  Arms: Tailored Therapy
Drug: Alectinib — TT arm
  Arms: Tailored Therapy
Drug: Brigatinib — TT arm
  Arms: Tailored Therapy
Drug: Palbociclib — TT arm
  Arms: Tailored Therapy
Drug: Ponatinib — TT arm
  Arms: Tailored Therapy
Drug: Vismogedib — TT arm
  Arms: Tailored Therapy
Drug: Itacitinib — TT arm
  Arms: Tailored Therapy
Drug: Ipatasertib — TT arm
  Arms: Tailored Therapy
Drug: Entrectinib — TT arm
  Arms: Tailored Therapy
Drug: Atezolizumab — TT arm
  Arms: Tailored Therapy
Drug: Nivolumab — TT arm
  Arms: Tailored Therapy
Drug: Ipilimumab — TT arm
  Arms: Tailored Therapy
Drug: Pemigatinib — TT arm
  Arms: Tailored Therapy
Drug: Oncology Drugs — Standard of Care Arm
  Arms: Standard of Care
Drug: Pralsetinib — TT arm
  Arms: Tailored Therapy
Drug: Selpercatinib — TT arm
  Arms: Tailored Therapy
Drug: Talazoparib — TT arm
  Arms: Tailored Therapy
Drug: Tepotinib — TT arm
  Arms: Tailored Therapy
Drug: Alpelisib — TT arm
  Arms: Tailored Therapy

SUMMARY:
This is a randomized, prospective, multicenter, Proof of Concept, Phase II clinical trial Study. The main objective of the study is to evaluate the efficacy (meant as overall response rate ORR) of TT (targeted Therapy) vs SoC (standard of Care) in patients with progressive disease (recurrent and/or metastatic) of breast cancer, metastatic gastro-intestinal tumors, non small cell lung cancer (NSCLC) or others. Patients should have completed at least 1 line of treatment and no more than 2 as defined by the current version of the AIOM (Italian Association of Medical Oncology) guidelines. Patients are included if surgery is contraindicated.

DETAILED DESCRIPTION:
Personalizing cancer medicine depends on the implementation of personalized diagnostics and therapeutics. Detailed genomic and gene expression signatures screening are likely to play a central role in this. Personalized Medicine has been widely depicted as a striking innovation, that is able to reform the standard approach to disease management, replacing the one-size-fits-all scheme of medicine with a single-patient-sized medical intervention.

Personalized medicine promoters usually highlight its potential to combine a more effective health-care with costs containment, according to the following rules:

* monitoring of disease risks and more effective prevention;
* early intervention;
* selection of optimal therapy;
* reduction of trial-and-error prescribing and reduction of adverse drug reactions;
* exclusion of unnecessary drugs;
* therapeutic drug monitoring and disease progression/remission monitoring;
* increased patient compliance with therapy. In spite of expectations, many unsolved practical issues, from technical and scientific to ethical, legal and economic topics, are slowing down the translation of personalized medicine principles into medical practice. Furthermore, wide adoption of personalized strategies also has to deal with the peculiar rules, policy and reimbursement system of each country.

Application of Personalized Medicine in the real world seems entangled by the unmet need to develop evidence-based guidelines.

The benefits of personalized medicine in routine clinical practice have firstly emerged in oncology. The power of precision medicine in the field of anticancer therapy resides in the possibility to characterize the genomic profile of both the disease (eg somatic mutations in the tumor tissue or blood sample) and the patient (eg the germinal genomic profile). The first piece of information allows stratification of patients in responder and non-responder to specific drugs, improving efficacy and avoiding wasting of expensive medications as biological drugs. Personalized medicine for cancer can be classified in:

* targeted therapy (which bloks the growth of cancer cells by interfering with specific molecular targets of cancer cells) or
* immunotherapy (which use the body'immune system to fight cancer cells by stimulating the immune system) Targeted therapy belongs to Personalized Medicine approach and the study of genetic mutations on tumor tissue or blood sample (CTC or cfDNA ) are changing the scenario of the treatment approach of cancer patients.

In clinical practice, the use of target therapies driven by mutation's assessment has radically changed the survival of patients affected by breast cancer, NSCLC, melanoma, colo-rectal cancer, while the clinical application of specific gene expression signatures is driving the choice of the best adjuvant strategy in early breast cancer.

Despite the efficacy of such approach its use is restricted to a relatively small fraction of patients and the evaluation of mutation is conditioned by the primary site of the cancer, i.e. by the tumor histology. The current biological understanding leads to hypothesize that the cancer behavior is highly dependent from the underlying driver genetic alterations independently from the histology. It's widely demonstrated that such molecular alterations are detected regardless of the histology, and this has already modified the treatment approach of some cancers.

Furthermore, several studies have demonstrated the efficacy of the choice of treatment according to genomic evaluation regardless of its histology with acceptable cost-effectiveness profile.

In the context of precision medicine the Immuno-oncology is becoming Precision Immuno-oncology and the efforts of science are directed towards the identification of predictive biomarkers of response to immune checkpoint inhibitors.

Promising biomarkers are Microsatellite Instability (MSI) and the tumour mutational load (TMB). In particular TMB is a quantitative biomarker that reflects the total number of mutations carried by tumor cells. TMB is well-known to reflect neoantigens burden potentially recognized by the immune system. This has been shown to correlate with better anti-PD-1 response in particular for both pembrolizumab and nivolumab combined with ipilimumab .

The same findings were demonstrated in the OAK study considering peripheral blood mutational load and response to atezolizumab.

High tumor mutation burden (defined as tumors that have high ≥10 mutations/megabase, mut/mb) allows to identify 45% of patients who can benefit from immunotherapy regardless of PD-L1 expression. So, ever keeping in mind that although many evidences are available, the relationship between histology and genomic alterations is still under definition, as well as the relationship between the latter and gene expression.

The aim of the present investigation is to combine all of the information available to drive the therapy selection according to the genomic alteration profile. Therefore, the main objective of our study is to evaluate the efficacy of therapy according to genomic profile (TT - Tailored Treatment) versus Standard of Care (SoC). A molecular profile of the cancer will be evaluated on tumor tissue biopsy (using the Foundation One (with updated gene panel 324 gene reflecting CDx) at the time of patient inclusion in the trial and on circulating DNA fragments (i.e. using FoundationOne Liquid test) at the time of patient inclusion in the trial and at progression of disease.

This study is a Phase II, randomized, multicenter, Proof of Concept, clinical trial. Patients with progressive disease (recurrent and/or metastatic) of breast cancer, metastatic gastro-intestinal tumors, non small cell lung cancer (NSCLC) or others will be included. Patients should have completed at least 1 line of treatment and no more than 2 as defined by the current version of the AIOM guidelines. Patients are included if surgery is contraindicated.

Patients could have received targeted therapy for metastatic disease. A molecular profile of the cancer will be evaluated on tumor tissue biopsy and on ctDNA of around 1280 patients at patient inclusion.

After FO evaluations patients with actionable mutations, not previous identified with other methods, for which approved drugs according to histotype are available, will be excluded.

Once identified molecular abnormalities (not only those that are disease-specific), that can be modulated with target or immunotherapeutic intervention available within the present study, patients will be randomized to receive:

ARM A: Therapy at choice of physician, according to Standard of Care (SoC) ARM B: Tailored treatment according to genomic profile (Tailored Treatment, TT)

The Molecular Tumor Board (MTB) will define the target therapy and immunotherapy while standard treatment will be decided by study physicians.

Patients should remain in the treatment phase of the study until investigator assesses radiographic or clinical progressive disease, unmanageable toxicity, or study termination.

Tumor assessments will be conducted every 12 weeks from the date of randomization until any of the above events occurs.

Delays in treatment administration will not impact the timing of the tumor assessments. If a tumor assessment must be performed early/late, subsequent assessments will be conducted according to the original schedule of every 12 weeks from the date of randomization.

At the time of the first progression of disease:

* blood sample will be collected to evaluate the molecular profile of the cancer on circulating DNA fragments (i.e. using FoundationOne Liquid test)
* Study treatment (SoC or TT) will be interrupted waiting for the evaluations for the Rescue/Switched Phase

Tumor assessments must be conducted until progressive disease (PD for RECIST 1.1 or iCPD for iRECIST if clinically indicated), even if treatment has been discontinued due to investigator-determined PD or unacceptable toxicity.

After discontinuation of study treatment for reason different from progressive disease and withdrawal of consent, tumor assessments will continue until progression.

In addition, patients will be followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 at time of signing Informed Consent Form
2. Patients able and willing to provide a written informed consent to participate to the study
3. Patients with recurrent/metastatic breast, gastrointestinal cancer,non small cell lung cancer or others
4. Patients not treatable with potentially curative surgery ot other loco-regional treatments.
5. Patients should have been completed at least or failed the first line of treatment for breast cancer, gastro-intestinal, non small cell lung cancer or other cancer
6. ECOG performance status from 0 to 1
7. Molecular target not actionable with approved drugs identified during screening by profiling with FoundationOne CDX on biopsy and FoundationOne Liquid CDx on blood
8. Biopsiable disease (tumor biopsy mandatory for tumor profiling). The biopsy must be performed during the screening period, when patients complete the conventional therapy for their recurrent/metastatic cancer. Historical samples will be considered for the study if collected within 3 months before the ICF signature of the patient. Samples older than 3 months, with a maximum timeframe of 6 months, and collected before progression of disease after the last treatment administered will be considered upon clinical judgement of the Investigator, after confirmation by the coordinating site or MTB. Samples obtained from a biospy of a metastatic lesion in progression after the last treatment administered represent the optimal tissue sample for genomic testing. Patients with glioblastomas and high grade malignant gliomas can be enrolled with the historical tissue samples.
9. Measurable disease, eligible to standard treatment. Patients must have measurable or evaluable disease defined, per RECIST 1.1 or irCS (immune related Response Criteria), as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral computed tomography (CT) scan, Magnetic Resonance Imaging (MRI), or a subcutaneous or superficial lesion that can be measured with calipers by clinical exam. For lymph nodes, the short axis must be ≥15 mm. Patients who have assessable disease by physical or radiographic examination but do not fully meet the above definitions of measurable disease (but still remains measurable) are eligible and will be considered to have evaluable disease. Patient's whose disease cannot be objectively measured by physical or radiographic examination (e.g., elevated serum tumor marker only) are NOT eligible. PET scan could be performed, if clinically indicated. For PET response evaluation PERCIST criteria will be applied.
10. Adequate renal function defined by a serum creatinine <1.5xUNL (upper normal limit).
11. Adequate liver function test defined by SGOT & SGPT <3xUNL (5xUNL in case of liver metastases), and bilirubin level <1.5xUNL
12. Adequate bone marrow function defined by platelets >100,000/mm3, hemoglobin >10 g/dL, and neutrophils >1,000/mm3
13. For female of child-bearing potential and for all women < 1 years after the onset of menopause: a negative pregnancy test <72 hours before starting study treatment is required. If sexually active, female of childbearing potential must use "highly effective" methods of contraception for the study duration. Contraception should continue after the last treatment for 3 months or for longer periods according to what reported in the Appendix 1 of the Protocol
14. For male of reproductive potential: any sexually active male patient must use a condom while on study treatment. Contraception should continue after the last treatment for 3 months or for longer periods according to what reported in the Appendix 1 of the Protocol.

Exclusion Criteria:

1. Patients who have only bone and/or brain metastases
2. Patients treated with more than 2 lines for breast cancer, gastro-intestinal, non small cell lung cancer and other cancer
3. Patients with uncontrolled disease (untreated and/or sintomatic) and patients whose brain metastases have not been monitored for >2 months
4. Patients with well-established actionable targets for which approved and marketed targeted drugs are available (i.e. lung cancer with EGFR mutation, or ALK translocation, B-RAF mutant melanoma, GIST with KIT mutations or breast cancer with HER2 amplification)
5. Patient participating in another clinical trial with an experimental drug
6. Anticoagulation with anti-vitamin K (Low Molecular Weight Heparin [LMWH] is allowed)
7. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including uncontrolled diabetes, cardiac disease, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within one year, chronic liver or renal disease, active gastrointestinal tract ulceration, severely impaired lung function
8. Pregnant and/or breastfeeding women
9. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
10. HIV, HBV, or HCV infection as per specific test performed at the screening visit or known as per Medical History
11. Patients with documented contraindication to any of the IMPs that will be used for the study, as reported in the respective SmPcs/IBs and in Appendix 2
12. Patients treated with the following drugs, because of the risk of immunosuppression: Chronic or high-dose oral corticosteroid therapy, TNF-inhibitors and Anti-T cell antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
OVERALL RESPONSE RATE (ORR) | 42 months
  Evaluation of the ORR of the Treatment at choice of physicians, according to Standard of Care (SoC) or of the Tailored Treatment (TT).
  The ORR will be constructed according to the specific design of the study, therefore including also the Rescue Therapy Phase data.
  This means that the ORR will take into account 3 evaluations:
  * on the original final population ( i.e 384 patients divided into the 4 groups of type of cancer)
  * on the TT patients, which will include the original randomized TT patients and the patients switched from the standard of care therapy (SoC therapy) to the TT Therapy, this latter within the Rescue Therapy Phase (patients switching upon the first documented progression)
  * on the population composed by the original TT patients, the original SoC patients and the switched TT patients. This means that the total population analyzed will include the original 384 population data (as per randomization) and the additional switched TT patients.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) of SoC vs TT | 42 months
Time to Treatment Failure (TTF) of SoC vs TT | 42 months
Time to Next Treatment (TTNT) of SoC vs TT | 42 months
Concordance between molecular profile on tumor tissue and ctDNA | 42 months
  Will be evaluated the concordance between Foundation One results on tumor tissue and blood sample. Overlapping mutational results will be considered as "concordant" otherwise will be considered as "discordant". Both qualitative and quantitative differences in mutational status will be considered.
QoLs included in the two arms of the study of SoC vs TT | 42 months
  The QoL score will be measured in the two arms of the study (SoC and TT), using the EORTC QLQ-C30, a validated questionnaire designed to assess different aspects of health and quality of life for cancer patients. Data from the two Quality of Life (QoL) questionnaires will be descriptively analyzed.
The safety profile between the two treatment arms of SoC vs TT | 42 months
  Percentage of Participants with Adverse Events (AEs) or Serious AEs (SAEs).
Overall survival (OS) | 42 months
  ● Overall survival (OS) is defined as the time from randomization to death from any cause. Data for patients with no record of death will be censored at the last date they were known to be alive. The analysis of OS will follow the same methodology as the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Marchetti, Study Chair — Fondazione per la Medicina Personalizzata; Andrea Botticelli, Principal Investigator — Università degli Studi di Roma Sapienza
Locations (37):
- Italy (37):
  - OSPEDALI RIUNITI di ANCONA, Ancona
  - Centro Riferimento Oncologico, Aviano
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii - Bari, Bari
  - Asst Papa Giovanni Xxiii, Bergamo
  - Ospedale Bellaria, Bologna
  - Ospedale di Carpi, Carpi
  - Arnas Garibaldi- Nuovo Ospedale Garibaldi - Nesima, Catania
  - A.O. Mater Domini Catanzaro, Catanzaro
  - Azienda Ospedaliero-Universitaria Di Ferrara, Ferrara
  - E.O. Ospedali Galliera, Genova
  - Ospedale Policlinico San Martino, Genova
  - Ospedale Della Misericordia, Grosseto
  - I.R.S.T. Srl Irccs, Meldola
  - Ao Papardo, Messina
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Tumori Di Napoli Irccs Pascale, Napoli
  - Ospedale Classificato Sacro Cuore - Don Calabria, Negrar
  - I.R.C.C.S. Istituto Oncologico Veneto, Padua
  - Az.Osp.Univ.P.Giaccone, Palermo
  - Azienda Ospedaliera Di Perugia, Perugia
  - Casa Di Cura Privata Osp. P. Pederzoli, Peschiera del Garda
  - Azienda Usl Di Piacenza, Piacenza
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Nuovo Ospedale Di Prato - S. Stefano, Prato
  - Ospedale "Santa Maria Delle Croci", Ravenna
  - Arcispedale Santa Maria Nuova Di Reggio Emilia, Reggio Emilia
  - Az. Osp. Uni. Policlinico Umberto I, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Istituti Fisioterapici Ospitalieri- Ifo - Istituto Regina Elena, Roma
  - Ospedale Fatebenefratelli, Roma
  - Policl. Univ. Campus Bio Medico, Roma
  - Casa Sollievo della Sofferenza - Opera Padre Pio, San Giovanni Rotondo
  - Azienda Ospedaliera 'S. Maria' - Terni, Terni
  - AO Ordine Mauriziano, Torino
  - Humanitas Gradenigo, Torino
  - IRCCS Candiolo, Torino
  - Complesso Ospedaliero Di Belcolle- Ospedale Di Belcolle, Viterbo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marchetti P, Curigliano G, Biffoni M, Lonardi S, Scagnoli S, Fornaro L, Guarneri V, De Giorgi U, Ascierto PA, Blandino G, D'Amati G, Aglietta M, Cremolini C, Conte P, Crimini E, Ceracchi M, Pisegna S, Verkhovskaia S, Bordonaro R, Bracarda S, Butturini G, Del Mastro L, DeCensi A, Fabbri A, Fenocchio E, Gori S, Metro G, Pessino A, Pozzessere D, Puglisi F, Tamberi S, Zambelli A, Marino D, Capoluongo E, Cappuzzo F, Cerbelli B, Giannini G, Malapelle U, Mazzuca F, Nuti M, Pruneri G, Simmaco M, Strigari L, Tonini G, Martini N, Botticelli A; ROME trial investigators consortia. Genomically matched therapy in advanced solid tumors: the randomized phase 2 ROME trial. Nat Med. 2025 Oct;31(10):3514-3523. doi: 10.1038/s41591-025-03918-x. Epub 2025 Sep 29. PMID 41023484